CLINICAL TRIAL: NCT00354640
Title: A Trial Assessing the Effect of Simvastatin on the Pharmacokinetics of Anastrozole
Brief Title: Simvastatin and Anastrozole in Treating Postmenopausal Women With Ductal Carcinoma In Situ or Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J05100, CDR0000485361; P30CA006973 (NIH); JHOC-J05100 (Other: SKCCC); JHOC-SKCCC-J05100 (Other: SKCCC)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast cancer in situ; ductal breast carcinoma in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Anastrozole; Simvastatin; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anastrozole and Simvastatin (Experimental): This is a pharmacological study for women on anastrozole as adjuvant therapy for breast cancer to receive concurrent simvastatin for up to 14 days.
  Interventions: Drug: anastrozole; Drug: simvastatin; Other: pharmacological study; Procedure: adjuvant therapy

INTERVENTIONS:
Drug: anastrozole — 1 milligram tablet PO QD for 14 days
  Other Names: Arimidex
Drug: simvastatin — 40 milligram tablet PO QD for 14 days
  Other Names: Zocor
Other: pharmacological study — laboratory analysis
Procedure: adjuvant therapy — laboratory analysis

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of simvastatin and anastrozole may stop cancer from forming, growing, or coming back in patients with invasive breast cancer, ductal carcinoma in situ, or a high risk of breast cancer.

PURPOSE: This phase II trial is studying how well giving simvastatin together with anastrozole works in treating postmenopausal women with invasive breast cancer, ductal carcinoma in situ, or a high risk of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the effects of concurrent anastrozole and simvastatin on anastrozole's steady-state concentration in postmenopausal women with history of invasive breast cancer or ductal carcinoma in situ or at high risk for developing breast cancer.

Secondary

* Study the effect of concurrent simvastatin and anastrozole on estrogen suppression in these patients.

OUTLINE: This is a pilot study.

Patients continue to receive oral anastrozole once daily (as prior to study entry). They also receive oral simvastatin once daily for 14-18 days in the absence of unacceptable toxicity or diagnosis of new or recurrent breast cancer.

Patients undergo blood sample collection at baseline and after study therapy for analysis of anastrozole and hormone (estradiol and estrogen) concentrations.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets any of the following criteria:

  * History of invasive breast cancer
  * History of ductal carcinoma in situ
  * At high risk for breast cancer, defined as being on anastrozole for chemoprevention of breast cancer
* Receiving anastrozole for ≥ 30 days as adjuvant breast cancer treatment or for prevention of breast cancer
* No active breast cancer with known metastatic involvement
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* ECOG performance status 0-2
* AST and ALT ≤ 3 times upper limit of normal
* Creatinine clearance ≥ 30 mL/min
* No active liver disease
* No prior hypersensitivity to any HMG-CoA reductase inhibitor or any of its components
* No daily alcohol use of > 3 standard drinks/day

  * A standard drink is defined as 10 g of alcohol, which is equivalent to 285 mL of beer, 530 mL of light beer, 100 mL of wine, or 30 mL of liquor

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No cholesterol-lowering drug, including a statin, within the past 3 months
* No selective estrogen receptor modulator (SERM) within the past 3 months
* No other hormone therapy within the past 3 months
* No prior estrogen and/or progesterone hormone replacement therapy that lasted for ≥ 5 years

  * Vaginal estrogen preparations allowed
* No other concurrent statin or cholesterol-lowering drug
* No other concurrent SERM
* No other concurrent hormone therapy
* No other concurrent investigational drugs
* No concurrent CYP3A4 inhibitors, including itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, nefazodone, or cyclosporine
* No concurrent chemotherapy or biological agents
* No concurrent daily grapefruit juice > 8 oz/day
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven women were enrolled from December 2006 to September 2008.
Pre-assignment Details: Women were required to be taking anastrozole as adjuvant treatment for breast cancer.
Groups:
- Anastrozole and Simvastatin: adjuvant therapy : laboratory analysis
  pharmacological study : laboratory analysis
  simvastatin : 40 milligram tablet PO QD for 14 days
  anastrozole : 1 milligram tablet PO QD for 14 days
Period: Overall Study
Arm/Group | Anastrozole and Simvastatin
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anastrozole and Simvastatin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Concentrations
Description: The change in blood concentrations of anastrozole at baseline and 14 days was measured.
Time Frame: Baseline and 14 days
Population: Participants with blood samples for trough concentrations were included.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Anastrozole and Simvastatin
Number analyzed (Participants) | 9
ng/ml
  Anastrozole concentration | 4.2 [-6.2 to 22.1]
  Hydroxyanastrozole concentration | -0.03 [-0.14 to 0.08]

2. Secondary Outcome: Change in Serum Estradiol Levels
Description: The change in serum concentrations of estradiol at baseline and 14 days was measured.
Time Frame: Baseline and 14 days
Population: Participants with blood samples for trough concentrations were included.
Measure: Median (Full Range); unit: pmol/l
Arm/Group | Anastrozole and Simvastatin
Number analyzed (Participants) | 9
pmol/l | -3.0 [-19.0 to 9.5]

ADVERSE EVENTS:
Time Frame: 14 days
Description: Participants were assessed by a member of the study team at the end of simvastatin dosing.
Arm/Group | Anastrozole and Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Small sample size, difficulty in recruiting due to women either already taking a statin or on a different aromatase inhibitor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No